CLINICAL TRIAL: NCT02714972
Title: Reduction of Nocturnal Hypoglycemia and Hyperglycemia in the Home Using Predictive Algorithms, Pump Suspension, and Insulin Dosing in Children and Young Adolescents (PHM3)
Brief Title: Reduction of Nocturnal Hypoglycemia and Hyperglycemia in the Home Using Predictive Algorithms, Pump Suspension, and Insulin Dosing in Children and Young Adolescents
Acronym: PHM3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PHM3
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes; Hypoglycemia; Hyperglycemia; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects are randomized on a per-night level for when the PHHM will be active or not.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperglycemia Minimization Algorithm (Active Comparator): The hyperglycemia minimization algorithm will be running actively on the study laptop during the night and dose insulin if the algorithm predicts hyperglycemia. If hypoglycemia is predicted, the system will suspend the pump.
  Interventions: Device: Hyperglycemia Minimization Algorithm
- Predictive Low Glucose Suspend (No Intervention): The control algorithm will run passively and not dose additional insulin. If hypoglycemia is predicted, the system will suspend the pump.

INTERVENTIONS:
Device: Hyperglycemia Minimization Algorithm — The hyperglycemia minimization algorithm will be running actively on the study laptop during the night and dose insulin if the algorithm predicts hyperglycemia. If hypoglycemia is predicted, the system will suspend the pump.
  Arms: Hyperglycemia Minimization Algorithm

SUMMARY:
Objective: to gain experience in children and younger adolescents with in-home use of an algorithm that will dose insulin to minimize projected hyperglycemia overnight in addition to suspending the pump if hypoglycemia is projected overnight and to obtain feasibility, safety, and initial efficacy data

Study Design: randomized controlled trial, with randomization on a night level within subject Patient Population: Youth 6.0 - <15 years old with type 1 diabetes treated with daily insulin therapy for at least one year and an insulin infusion pump for at least 6 months who have HbA1c < 10.0%.

Sample Size: 30 subjects

Study Duration and Visit Schedule: duration approximately 3 months, with preliminary run-in activities followed by up to 90 days spent in clinical trial phase of study; clinic visits at enrollment, following CGM and system assessment run-in phases, at start of clinical trial phase, at 21-day point of clinical trial phase, and after 42 nights of successful system use

Major Efficacy Outcomes:

* Primary: time in range (70-180 mg/dl, 3.9-10.0 mmol/L) overnight.
* Secondary: time spent in hypoglycemia (<70 mg/dl, 3.9 mmol/L) and time spent in hyperglycemia (>180 mg/dl, 10.0 mmol/L) overnight.

Major Safety Outcomes: CGM measures of hypo- and hyperglycemia, including morning blood glucose and mean overnight sensor glucose; adverse events including severe hypoglycemia and diabetic ketoacidosis

DETAILED DESCRIPTION:
Subjects who are eligible for the clinical trial initially will use a Veo insulin pump and Enlite CGM sensor at home for a minimum of 6 days/week over a 2-week period to verify that the subject is able to use the CGM and insert sensors.

The first 10 subjects enrolled will be 11 to <15 years of age and will participate in an Algorithm Assessment Phase of approximately 10 nights of system use each with PLGS and Hyper Minimization active. Results of the approximate 100 nights will be reviewed with the study DSMB to assess safety and determine whether any adjustments to the algorithm parameters are needed. If adjustments are needed, the Algorithm Assessment Phase will be repeated with the same age restriction, using the same 10 subjects if possible. If no adjustments are needed and the DSMB judges it safe to continue the study, enrollment will continue across the full 6 to <15 age range.

Subjects who enroll in the study after the completion of the Algorithm Assessment Phase will use the closed-loop system at home for 5 nights of system use each with PLGS and Hyper Minimization active to demonstrate their ability to use the system and submit study data to the Coordinating Center.

Subjects who successfully demonstrate their ability to use the system at home as described above will be eligible for the randomized trial phase. This phase consists of use of the full system in the home for approximately 42 nights:

* Each night the blood glucose level will be checked with the BG meter and used to perform a calibration of the CGM. This calibration must occur no more than 90 minutes prior to activation of the system. NOTE: Subjects will be instructed to calibrate the CGM per manufacturer guidelines.
* Then the system will be activated, linking the CGM and insulin pump to the computer at the bedside.
* A randomization schedule on the laptop will be used to determine whether the system will run in PLGS+Hyper Minimization mode or PLGS-only.

  * Subjects will be blinded as to whether the system is running in PLGS+Hyper Minimization mode or PLGS-only.
  * There will not be an alarm if the pump shuts off or if automated insulin dosing occurs. The CGM alarm will be set to 60 mg/dL (3.3 mmol/L). When a CGM alarm occurs, the subject will be asked to measure the blood glucose with a BG meter, if he/she is aware of the alarm.
  * The time period for outcome assessment each night will be from the time the system is activated until it is turned off in the morning.
  * Pump shut off, when it occurs, will be for up to 120 minutes in a 150-minute period, and no more than 180 minutes for the entire night. Multiple instances of pump suspension can occur if there are recurrent predictions of hypoglycemia during the night.
* Small correction boluses of insulin will be delivered when the system predicts that hyperglycemia above a pre-set threshold will occur, with insulin-on-board constraints and cumulative delivery limits to minimize the likelihood of excessive insulin delivery.
* Subjects will be asked to check blood glucose with the study BG meter each morning prior to breakfast and enter the results using the controller software interface. The subject will be instructed to contact the study physician if the morning blood glucose value is <60 mg/dl (3.3 mmol/L) or >300 mg/dl (16.7 mmol/L). Monitoring processes will ensure that the subject can be contacted if these values are not reported as required or are out of range.
* Subjects will be asked to record all overnight carbohydrate intake using the controller software interface.
* Subjects will be asked to perform periodic CGM data uploads using the controller software interface. Monitoring processes will ensure that the subject can be contacted if these uploads do not occur as required, or if review of an upload reveals any extreme, prolonged episodes of hypoglycemia or hyperglycemia, or elevated morning blood glucose values.

Once approximately 200 nights of randomized clinical trial phase data are available, the study DSMB will perform another data review to determine whether it is safe to continue the study. Subjects already using the study system at home will continue to use it during the DSMB review process, but no additional subjects will begin home use of the system until the DSMB review is complete.

Upon completion of the study, subjects as well as study clinicians will be asked to complete a human factors usability questionnaire regarding use of the study system.

There will be a follow-up (optional) extension phase for subjects who exhibit safe and competent use of the system at home. They may be given the option to continue home use of the system for up to 56 days to assess whether data-driven, subject-level customization of algorithm parameters improves glycemic outcomes compared with generic algorithm parameters that are identical for each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year and an insulin infusion pump for at least 6 months The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
2. Age 6.0 to <15.0 years
3. HbA1c < 10.0%

   * Measured with DCA2000 or equivalent device for assessing eligibility
   * HbA1c measurements performed as part of usual clinical care within 2 weeks prior to obtaining informed consent for participation in the trial may be used.
4. Uninterrupted internet access while study system is being used overnight and for upload of study data in the morning
5. Living with a family member/guardian ("companion") committed to participating in all study activities, and being present and available to provide assistance when the system is being used at night
6. An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

1. Diabetic ketoacidosis in the past 6 months
2. Hypoglycemic seizure or loss of consciousness in the past 6 months
3. History of seizure disorder (except for hypoglycemic seizure)
4. History of any heart disease including coronary artery disease, heart failure, or arrhythmias
5. Cystic fibrosis
6. Current use of oral/inhaled glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
7. History of ongoing renal disease (other than microalbuminuria). Creatinine level must have been obtained within the last year if subject has diabetes of >10 years duration. If creatinine is > 1.5 mg/dL (132 µmol/L), the subject is excluded.
8. Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

   * Inpatient psychiatric treatment in the past 6 months
   * Uncontrolled adrenal disorder
   * Abuse of alcohol
9. Pregnancy (Negative urine pregnancy test required for females who have experienced menarche as well as agreement from subject and parent/guardian to use a form of contraception to prevent pregnancy while participant is in the study. Subjects who become pregnant will be discontinued from the study)
10. Liver disease as defined by an ALT greater than 3 times the upper limit of normal

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Comparison of percent time in range overnight between the two treatment arms | Up to 42 nights
  A single percentage calculated for each subject by pooling all CGM readings from the PLSG+HM nights will be compared with the corresponding percentage obtained by pooling all of the data from PLGS-only nights for the same subject. All CGM readings regardless of the amount of data will be weighted equally in the pooled percentage regardless of how they distribute across nights.

SECONDARY OUTCOMES:
Mean overnight sensor glucose | Up to 42 nights
Glucose standard deviation and coefficient of variation | Up to 42 nights
Percent of sensor measurements below 50 mg/dl (2.8 mmol/L) | Up to 42 nights
Percent of sensor measurements below 60 mg/dl (3.3 mmol/L) | Up to 42 nights
Percent of sensor measurements below 70 mg/dl (3.9 mmol/L) | Up to 42 nights
Area under the curve 70 mg/dl (3.9 mmol/L) | Up to 42 nights
Low blood glucose index | Up to 42 nights
Percent of sensor measurements above 180 mg/dl (10.0 mmol/L) | Up to 42 nights
Percent of sensor measurements above 250 mg/dl (13.9 mmol/L) | Up to 42 nights
Percent of sensor measurements above 300 mg/dl (16.7 mmol/L) | Up to 42 nights
Area under the curve 180 mg/dl (10.0 mmol/L) | Up to 42 nights
High blood glucose index | Up to 42 nights
Percent of sensor measurements between 70 mg/dl (3.9 mmol/L) | Up to 42 nights
Percent of sensor measurements between 140 mg/dl (7.8 mmol/L) | Up to 42 nights
Percentage of nights with events of sensor glucose below 50 mg/dl (2.8 mmol/L), 60 mg/dl (3.3 mmol/L), and 70 mg/dl (3.9 mmol/L) continuously for more than 0, 10, 25, 30, 60, and 120 minutes | Up to 42 nights
Percentage of nights with events of sensor glucose below 50 mg/dl (2.8 mmol/L), 60 mg/dl (3.3 mmol/L), and 70 mg/dl (3.9 mmol/L) cumulatively for more than 30, 60, 120, and 180 minutes | Up to 42 nights
Percentage of nights with events of sensor glucose above 180 mg/dl (10.0 mmol/L), 250 mg/dl (13.9 mmol/L), and 300 mg/dl (16.7 mmol/L) continuously for more than 0, 30, 60, and 120 minutes | Up to 42 nights
Percentage of nights with events of sensor glucose above 180 mg/dl (10.0 mmol/L), 250 mg/dl (13.9 mmol/L), and 300 mg/dl (16.7 mmol/L) cumulatively for more than 60, 120, and 180 minutes | Up to 42 nights
Mean morning blood glucose (subject-level data) and percent of morning with blood glucose below 50 mg/dl (2.8 mmol/L), 60 mg/dl (3.3 mmol/L), 70 mg/dl (3.9 mmol/L) (night-level data) | Up to 42 nights
Mean morning blood glucose (subject-level data) and percent of morning with blood glucose between 70 mg/dl (3.9 mmol/L) and 180 mg/dl (10.0 mmol/L) (night-level data) | Up to 42 nights
Mean morning blood glucose (subject-level data) and percent of morning with blood glucose above 180 mg/dl (10.0 mmol/L), 250 mg/dl (13.9 mmol/L), and 300 mg/dl (16.7 mmol/L) (night-level data) | Up to 42 nights
Amount of total (manual, automatic, combined) and insulin boluses | Up to 42 nights

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Buckingham, MD, Study Chair — Stanford University; John W Lum, MS, Study Director — Jaeb Center for Health Research; Roy Beck, MD, PhD, Principal Investigator — Jaeb Center for Health Research
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado